CLINICAL TRIAL: NCT05083130
Title: Evaluation of Awake Prone Positioning Effectiveness in Moderate to Severe COVID-19
Brief Title: Awake Prone Positioning in Moderate to Severe COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06NV
Record Dates: First submitted 2021-10-10; First posted 2021-10-19 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: COVID-19; SARS-CoV2 Infection; COVID-19 Acute Respiratory Distress Syndrome; Acute Hypoxemic Respiratory Failure; Respiratory Distress Syndrome, Adult
Keywords: prone position; severe COVID-19; acute respiratory distress syndrome (ARDS); Vietnam
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Open label randomised controlled trial comparing standard care to prone position
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (No Intervention): Standard care will consist of routine clinical care, including any advice to lie in prone position as routinely recommended by participating sites
- prone position (Experimental): prone position group will have a special intervention team who visits patients' rooms aiming for patients to maintain the prone position for at least 8 hours a day
  Interventions: Behavioral: a wake prone positioning

INTERVENTIONS:
Behavioral: a wake prone positioning — The team will give written and verbal advice and if necessary aid patients' positioning themselves in the prone position for at least 8 hours per day. The exact duration of prone sessions will be determined according to ward schedules to take account of nursing procedures, meal times and mitigation strategies. Other methods to encourage the maintenance of prone position includes phone calls to patients, carers or education of carers.
  Arms: prone position

SUMMARY:
The purpose of this study is comparing vital signs between standard care and prone position groups. Standard care will consist of routine clinical care, including any advice to lie in prone position as routinely recommended by participating sites. For those randomized to prone position, a special intervention team will visit patients' rooms aiming for patients to maintain the prone position for at least 8 hours a day.

DETAILED DESCRIPTION:
This study is a pragmatic open label randomised controlled trial. After being informed about the study and potential risks, all patients having written informed consents will be randomised into two groups. Standard care group will consist of routine clinical care, including any advice to lie in prone position as routinely recommended by participating sites. To reduce bias, the study team will make visits at a similar schedule to those to patients in the intervention group, however these visits will be confined to general advice and measurement of vital signs. Patients will receive written advice more general in nature about COVID-19 disease. For those randomized to prone position group, a special intervention team will visit patients' rooms aiming for patients to maintain the prone position for at least 8 hours a day. The team will give written and verbal advice and if necessary aid patients' positioning themselves in the prone position. The exact duration of prone sessions will be determined according to ward schedules to take account of nursing procedures, meal times and mitigation strategies. Other methods to encourage the maintenance of prone position includes phone calls to patients, carers or education of carers. Compliance with the intervention will be evaluated by observation (manual and using in-room cameras) at fixed time intervals. In a subgroup of 100 patients accelerometer/gyrometer devices will be used to measure movement and position (this will be expanded to all patients if equipment is available). Other outcome measures (SpO2, heart rate etc) will be measured using standard monitoring equipment currently used at study sites, including wearable devices.

ELIGIBILITY:
Inclusion Criteria:

* Probable or confirmed COVID-19 infection according to WHO criteria
* Moderate or severe COVID-19 respiratory infection according to Vietnamese guidelines
* Requirement for supplemental oxygen therapy

Exclusion Criteria:

* Invasive mechanical ventilation, or non-invasive ventilation (NIV) with CPAP or BiPAP or imminent need for these
* Contraindications to prone position (see Appendix 5)
* Pregnancy
* Severe obesity (BMI >35),
* Altered level of consciousness (GCS <13)
* Attending doctor judged prone position to be unsuitable for the patient for any reason
* Patients in whom there is a decision that care will not be escalated
* Failure to have informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who require escalation of respiratory therapy | Up to 28 days after enrollment
  Escalation of respiratory therapy within 28 days of randomization, defined as any of the following:
  * Escalation to next level respiratory support (with lowest level nasal cannula or face mask, escalating through HFNC to NIV or mechanical ventilation).
  * Intubation

SECONDARY OUTCOMES:
Fatal event | Up to 28 days after enrollment
  all-cause of death within first 28 days will be compared between groups
Duration of hospital stay | Up to 2 months after enrollment
  Days since admission to discharge
Improvement in oxygen related parameters | Up to 28 days after enrollment
  SpO2, respiratory rate, heart rate, FiO2, ROX index will be documented before and at end of period of prone positioning every day. The improvement will be measured by resolution of them compared with baseline parameters
Number of adverse events | Up to 28 days after enrollment
  An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. The severity of all AEs in this trial should be graded in line with the toxicity grading in Toxicity grading and management (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Louise C Thwaites, MD. PhD., Principal Investigator — University of Oxford, UK
Locations (1):
- Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data of this study may be requested for publication by journals. Sharing anonymised data with future similar/suitable studies will be decided by the sponsor, PIs and the authority agency where the data was collected. No identifiable information will be shared with any other person/organisation
Supporting Information: Study Protocol

REFERENCES:
- [Background] Dondorp AM, Hayat M, Aryal D, Beane A, Schultz MJ. Respiratory Support in COVID-19 Patients, with a Focus on Resource-Limited Settings. Am J Trop Med Hyg. 2020 Jun;102(6):1191-1197. doi: 10.4269/ajtmh.20-0283. PMID 32319424
- [Background] Gonzalez-Seguel F, Pinto-Concha JJ, Aranis N, Leppe J. Adverse Events of Prone Positioning in Mechanically Ventilated Adults With ARDS. Respir Care. 2021 Dec;66(12):1898-1911. doi: 10.4187/respcare.09194. Epub 2021 Jul 23. PMID 34301802
- [Background] Ehrmann S, Li J, Ibarra-Estrada M, Perez Y, Pavlov I, McNicholas B, Roca O, Mirza S, Vines D, Garcia-Salcido R, Aguirre-Avalos G, Trump MW, Nay MA, Dellamonica J, Nseir S, Mogri I, Cosgrave D, Jayaraman D, Masclans JR, Laffey JG, Tavernier E; Awake Prone Positioning Meta-Trial Group. Awake prone positioning for COVID-19 acute hypoxaemic respiratory failure: a randomised, controlled, multinational, open-label meta-trial. Lancet Respir Med. 2021 Dec;9(12):1387-1395. doi: 10.1016/S2213-2600(21)00356-8. Epub 2021 Aug 20. PMID 34425070
- [Derived] Phong NT, Duc DH, Hai HB, Nguyen NT, Khoa LDV, Khanh LTT, Tran LHB, Linh NTM, Van CTC, Thao DP, Trinh NTD, Kieu PT, Truong NT, Hoang VT, Ngoc NT, Vien TTD, Ly VT, Khoa TD, Beane A, Anibal J; OUCRU COVID RESEACH GROUP; Thwaites GE, Geskus R, Clifton D, Dung NTP, Kestelyn E, Glover G, Tan LV, Yen LM, Tung NLN, Dung NT, Thwaites CL. Awake prone positioning effectiveness in moderate to severe COVID-19 a randomized controlled trial. Wellcome Open Res. 2024 Dec 7;9:543. doi: 10.12688/wellcomeopenres.22792.2. eCollection 2024. PMID 39654551
- See also: Prone position in ARDS patients: why, when, how and for whom. Intensive Care Med [Internet]. 2020;46(12):2385-96. — https://doi.org/10.1007/s00134-020-06306-w
- See also: Prone positioning in severe acute respiratory distress syndrome. N Engl J Med [Internet]. 2013 Jun 6 [cited 2014 May 23];368(23):2159-68 — http://www.ncbi.nlm.nih.gov/pubmed/23688302
- See also: Vietnam Ministry of Health guideline on COVID-19 management, treatment — https://kcb.vn/quyet-dinh-so-4689-qd-byt-ngay-06-10-2021-huong-dan-chan-doan-va-dieu-tri-covid-19-cap-nhat-lan-thu-7.html
- See also: Effect of awake prone position on diaphragmatic thickening fraction in patients assisted by noninvasive ventilation for hypoxemic acute respiratory failure related to novel coron — https://doi.org/10.1186/s13054-021-03735-x
- See also: Effect of early awake prone positioning application on prognosis in patients with acute respiratory failure due to COVID-19 pneumonia: a retrospective observational study. Brazilian J Anesthe — https://doi.org/10.1016/j.bjane.2021.07.029
- See also: Expert consensus statements for the management of COVID-19-related acute respiratory failure using a Delphi method. Crit Care [Internet] — https://doi.org/10.1186/s13054-021-03491-y